CLINICAL TRIAL: NCT03382470
Title: Partnership to Enhance Antimicrobial Use in Resource-Limited Settings (PEARL): An Assessment of Need and Feasibility of Antimicrobial Stewardship Programs
Brief Title: Impact of Antimicrobial Stewardship Programs in the Global Setting
Acronym: PEARL
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Moi University (Other); Kilimanjaro Christian Medical Centre, Tanzania (Other); Ruhuna University, Sri Lanka (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00089077
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Resistance Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Antimicrobial stewardship advice — A basic antimicrobial stewardship team will be created at each site. The team will provide advice on the treatment of urinary tract infections and asymptomatic bacteriuria during the second half of the study.

SUMMARY:
Antimicrobial resistance is one of the greatest threats to human health, and is driven by inappropriate antimicrobial use. Antimicrobial stewardship programs (ASPs) improve the use of antimicrobials in hospitals. The purpose of this study is to identify the need for and barriers to implementation of ASPs in three hospitals in Sri Lanka, Kenya, and Tanzania.

DETAILED DESCRIPTION:
Antimicrobial resistance is one of the greatest threats to human health, and is driven by the inappropriate antimicrobial use. Antimicrobial stewardship programs (ASPs) improve the use of antimicrobials. The purpose of this study is to identify the need for and barriers to implementation of ASPs in three hospitals in Sri Lanka, Kenya, and Tanzania. The impact of creating a basic ASP will be assessed at each hospital.

ELIGIBILITY:
Inclusion Criteria: All patients admitted to the medical wards -

Exclusion Criteria: None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the adult medical wards at the three hospitals during the duration of the study will be eligible.
Sampling Method: Probability Sample
Enrollment: 3115 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Appropriate antimicrobial use, for example for urinary syndromes | 6 months
  A composite outcome will be created for 'inappropriate' antibiotic use. This outcome will consist of 1) Unnecessary treatment for asymptomatic bacteriuria, 2) Inappropriate duration of therapy for urinary tract infection (UTI)/ cystitis/ pyelonephritis (binary outcome- yes/no), and 3) Unnecessary double coverage for UTI/ cystitis/ pyelonephritis (binary outcome- yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Gayani Tillekeratne, MD MSc, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Teaching Hospital Karapitiya, Galle, Sri Lanka

IPD SHARING:
Plan to Share IPD: No